CLINICAL TRIAL: NCT00002650
Title: PHASE II DOUBLE-BLIND CHEMOPREVENTION TRIAL OF HIGH DOSE FOLIC ACID VERSUS PLACEBO IN PATIENTS WITH RESECTED COLORECTAL POLYPS
Brief Title: High-Dose Folic Acid in Preventing Colorectal Cancer in Patients Who Have Had Polyps Surgically Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000064180; E-8292; NCI-P95-0066
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folic Acid

INTERVENTIONS:
Dietary Supplement: folic acid

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of folic acid may be an effective way to prevent colorectal cancer in patients with polyps that have been surgically removed.

PURPOSE: Randomized phase II trial to study the effectiveness of high-dose folic acid in preventing colorectal cancer in patients who have had polyps surgically removed within 18 months of the trial.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether high-dose folic acid decreases global DNA hypomethylation, as well as other intermediary markers, in normal-appearing colonic epithelium of patients with colonic adenomas. II. Determine whether a decrease in global DNA hypomethylation and other intermediary markers can be induced safely and whether these effects persist after folic acid is discontinued in these patients. III. Confirm pilot data that indicates patients with adenomas have widespread DNA hypomethylation of the colorectal mucosa compared to controls. IV. Evaluate the effect of folic acid on the clinical course and rate of recurrence of adenomatous polyps in these patients. V. Study a control group of patients with no history of neoplastic, hyperplastic, or inflammatory colorectal lesions.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and age (50-70 vs 30-49 and over 70). Patients with adenomatous polyps at least 10 mm at colonoscopy are randomized to 1 of 2 treatment arms. Patients found to have no neoplastic, hyperplastic, or inflammatory polyps at colonoscopy are assigned to a control (untreated) group and complete laboratory studies and a baseline food frequency questionnaire only. Arm I: Patients receive folic acid daily. Arm II: Patients receive placebo daily. Treatment continues in both arms for 1 year in the absence of unacceptable toxicity or disease progression. Patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 80 patients (30 per arm and 20 for the control group) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Colonic adenoma(s) of at least 10 mm completely resected within 18 months prior to randomization or suspected adenomatous polyp(s) Colonoscopy with submission of at least 7 rectosigmoid biopsies required at entry No benign hyperplastic polyps or polyps less than 10 mm to be eligible for treatment No polyposis coli (i.e., more than 100 polyps in colon) No history of invasive colorectal cancer

PATIENT CHARACTERISTICS: Age: 21 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count greater than 100,000/mm3 Hemoglobin greater than 10 g/dL No untreated pernicious anemia Hepatic: Bilirubin less than 2 mg/dL ALT less than 2 times normal Alkaline phosphatase less than 2 times normal PT normal Renal: Not specified Gastrointestinal: No intestinal malabsorption No inflammatory bowel disease Other: No seizure within the past year No poor medical risk No other malignancy within past 5 years except basal cell cancer, superficial skin cancer, or carcinoma in situ of the cervix No vitamin B12 deficiency (less than 200 pg/mL) Not pregnant or nursing Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent methotrexate Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics No prior small bowel resection Other: No concurrent anticonvulsants No concurrent drugs that markedly interfere with folate absorption or metabolism (e.g., sulfasalazine and phenytoin) No concurrent vitamins during and for 2 years after beginning of study

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1995-06-12 (Actual); Primary Completion 2004-10-17 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Mason, MD, Study Chair — Tufts Medical Center Cancer Center
Locations (8):
- United States (8):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts
  - USDA Human Nutrition Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin